CLINICAL TRIAL: NCT04958460
Title: Effect of Bifidobacterium Bifidum (Bf-688) on Clinical Characteristics and Gut Microbiota in Attention-deficit/Hyperactivity Disorder: a Double-blind Randomized-control Trial
Brief Title: Effect of Probiotics on ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wang Liang-Jen (Other)
Responsible Party: Sponsor-Investigator, Wang Liang-Jen, Professor and Visiting Staff, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201901479A3C601
Record Dates: First submitted 2021-04-23; First posted 2021-07-12 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: ADHD; Probiotics; Gut Microbiota; Psychiatry; Clinical Trial
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics group (Experimental): Probiotics
  Candidates conditions excluded:
  1. Patients with major mental or neurological diseases such as intellectual disability, autism group disorders, schizophrenia, severe depression, bipolar disorder, epilepsy, brain injury, etc.
  2. Those who have serious gastrointestinal diseases, physiological diseases or genetic diseases that will affect the results of intestinal microflora assessment
  3. Have received ADHD-related drug treatment (containing Methylphenidate or Atomoxetine) in the past month.
  4. Have used antibiotics or edible probiotic-related products (including drops, tablets, capsules, bacterial powder) in the past month.
  5. Participated in other clinical research in the past month.
  6. Vegetarians or those currently undergoing special diet therapy.
  7. Evaluation by the host is not suitable for entering the test.
  Interventions: Other: BF688
- Control group (Placebo Comparator): Placebo
  Candidates conditions excluded:
  1. Patients with major mental or neurological diseases such as intellectual disability, autism group disorders, schizophrenia, severe depression, bipolar disorder, epilepsy, brain injury, etc.
  2. Those who have serious gastrointestinal diseases, physiological diseases or genetic diseases that will affect the results of intestinal microflora assessment
  3. Have received ADHD-related drug treatment (containing Methylphenidate or Atomoxetine) in the past month.
  4. Have used antibiotics or edible probiotic-related products (including drops, tablets, capsules, bacterial powder) in the past month.
  5. Participated in other clinical research in the past month.
  6. Vegetarians or those currently undergoing special diet therapy.
  7. Evaluation by the host is not suitable for entering the test.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Administrated 1 packet of maltodextrin (as placebo of Bf-688) in the morning and evening
  Arms: Control group
Other: BF688 — Administrated 1 pack each morning and evening (5×109 CFUs per day)
  Arms: Probiotics group

SUMMARY:
Attention-Deficit/Hyperactivity Disorder (ADHD) is a common neurodevelopmental disorder. Gut microbiome dysbiosis may be associated with the pathophysiology of ADHD. Investigators previously found the relative abundance of Sutterella stercoricanis were increased and Bifidobacterium bifidum were decreased in the ADHD group. Investigators hypothesize that ADHD patients receiving supplementary Bifidobacterium bifidum (Bf-688) is able to increase the proportion of Bf-688; inhibit the proportion of Sutterella; and improve ADHD symptoms.

DETAILED DESCRIPTION:
Aims:

Investigators will conduct an open-label, single arm study and a randomized, double-blind clinical trial to examine whether Bf-688 can achieve similar effects to therapeutic drugs for ADHD.

Methods:

The duration of this clinical trial is expected to be 2 years (March 2020 to February 2022).

1. In the first stage of study, investigators will conduct an open-label, single arm study. Investigators will recruit 30 children aged 4-16 who are diagnosed as ADHD who are eligible to participate in the trial. The patients will be administrated with Bf-688, 1 pack each morning and evening (5×109 colony forming units (CFUs) per day) for 8 weeks. At the baseline, 2nd, 4th and 8th week, the clinical symptoms of ADHD will be evaluated using the SNAP-IV and ADHD-RS. At weeks 0 and 8, blood samples and fecal samples will be collected and psychological tests will be performed.
2. In the second stage of study, This clinical trial is a prospective, randomized, double-blind, parallel-controlled clinical trial for children aged 6-12 years old who are diagnosis of ADHD and who are currently receiving ADHD drug therapy. A total of 120 patients will be recruited in this trial. All subjects will be randomly assigned (allocation ratio 1:1) to one of the following two groups (60 people in each group):

(1) Probiotics group: The original ADHD drug will be continuously used, and the Bf-688 packet (5×109 CFUs) will be administrated in the morning and in the evening daily.

(2) Placebo group: The original ADHD drug will be continuously used, and the placebo packet will be administrated in the morning and in the evening daily.

The patients will take the above prescription for 12 consecutive weeks. At the 0th, 4th, 8th, and 12th weeks, parents and teachers will be asked to fill SNAP-IV, and the researcher will use ADHD-RS to evaluate the clinical symptoms of ADHD. At the 0th week and 12th week, stool samples will be collected and psychological tests will be performed (CPT and CATA). Nucleic acid sequencing technology is used to identify bacterial species in feces, and high-throughput 16S rRNA sequences can be quickly obtained through Next Generation Sequencing (NGS), and fecal metabolites analysis.

Expected results:

Investigators expect to find that Bf-688 exhibit significant better effects than the placebo group for treating ADHD patients. This result will validate that gut microbiota modification may be beneficial for the behavioral symptoms of ADHD children, and the outcome may have the potential for patent and commercialization.

ELIGIBILITY:
Inclusion Criteria:

* ADHD

Exclusion Criteria:

* Autism
* MR
* Developmental Delay
* Vegetarian

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Kiddie-Schedule for Affective Disorder and Schizophrenia-Epidemiological Ver- sion (K-SADS-E) | At the baseline
  screening
The Chinese version of Swanson, Nolan and Pelham IV Scale (SNAP-IV) | At the baseline
  ADHD
The Chinese version of Swanson, Nolan and Pelham IV Scale (SNAP-IV) | 2nd week
  ADHD
The Chinese version of Swanson, Nolan and Pelham IV Scale (SNAP-IV) | 4th week
  ADHD
The Chinese version of Swanson, Nolan and Pelham IV Scale (SNAP-IV) | 8th week
  ADHD

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Jen Wang, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Liang-Jen Wang, Kaohsiung City, Taiwan